CLINICAL TRIAL: NCT01920217
Title: Identification Sepsis Related SNP by Whole Exome Sequencing: a Prospective Observational Study
Brief Title: Identification Sepsis Related Single Nucleotide Polymorphism (SNP) by Whole Exome Sequencing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Huijuan Wang, Dr, Chinese PLA General Hospital
Other Study IDs: 301PLAGH20130610
Record Dates: First submitted 2013-08-08; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Sepsis
Keywords: sepsis; SNP; mortality
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — whole blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- normal control
- Sepsis group

SUMMARY:
Sepsis is a common cause of death in intensive care unit, timely and accurate diagnosis and treatment directly affect the survival rate. Single nucleotide polymorphism (SNP) was promising genetic biomarker for sepsis patients. The present study was designed to screen several SNP by whole exome sequencing which evaluate the sepsis related snp site in order to be a new target for the treatment of sepsis.

DETAILED DESCRIPTION:
The study is a non-intervention, prospective observational study. Purpose of this sudy is to screening several SNPs by whole exome sequencing which can be used as genetic marker for sepsis patients. We will collect whole blood samples from patients with sepsis inRespiratory Intensive Care Unit (RICU), the Emergency Intensive Care Unit (EICU), or the Department of Surgery's ICU 301 Hospital since January 2013, and then whole exome sequencing was used to Screen SNPs which were related to sepsis. Then another 500 sepsis patients and 500 normal controls were used to validated the sequencing results.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sepsis
* Patients who agree with the study

Exclusion Criteria:

* Aged <18 years;
* Into the group who died within 24 hours;
* Agranulocytosis (<0.5 × 109 / L);
* Combined HIV infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: within 24 hours after admited in ICU
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
sepsis related SNP site | 28 days after admitted to ICU

CONTACTS AND LOCATIONS:
Overall Officials: Huijuan Wang, Dr, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA general hospital, Beijing, Beijing Municipality, China